CLINICAL TRIAL: NCT04359563
Title: You.Mind! | Boosting First-line Mental Health Care for Youngsters Suffering From Chronic Conditions With Mindfulness: A Randomised Staggered Within-subjects Design
Brief Title: You.Mind! | Boosting First-line Mental Health Care for Youngsters Suffering From Chronic Conditions With Mindfulness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Fondation Huoshen (Unknown)
Responsible Party: Principal Investigator, Katleen Van der Gucht, Principal Investigator, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: S63485
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Chronic Illness
Keywords: Emotional Distress; Quality of Life
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The study uses a randomized staggered within-subjects design in which participants are randomized to a baseline assessment phase of 14 to 28 days duration. During the subsequent intervention phase, all participants receive an 8-week Mindfulness-Based Intervention. Participants complete daily (every 3 days during intervention and follow-up phases) experience sampling method (ESM) measurements throughout the baseline, intervention and follow-up phases. Before randomisation, directly post-intervention and at 3 months follow-up, participants complete self-report questionnaires and ESM measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Intervention (Experimental): The MBI programme adheres to a standardized protocol developed from MBSR (Kabat-Zinn, 1990) and MBCT (Segal et al., 2012) manuals and is adjusted to an adolescent population. Adjustments are based on the investigator's ample experience with mindfulness and adolescents in different contexts. Key objectives are: (1) to increase awareness of one's present moment experience; (2) to teach an attitude of openness and acceptance (non-judging) toward one's experience. This accepting attitude changes the person's relationship with the experience, being a detached and non-reactive orientation. Participants learn to recognize entanglement with one's thoughts and emotions and there is an increased understanding of one's spontaneous reactions. If adolescents adopt these skills, their negative emotions and cognitions will no longer be reinforced, creating the opportunity to deal with problematic thoughts and feelings.
  Interventions: Behavioral: Mindfulness-Based Intervention

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — The MBI consists of four 2h online group sessions spread over eight weeks. In between sessions, online support will be offered to assist participants in their practice. Each session consists of guided mindfulness exercises (e.g., focus on the breath, body scan, breathing space, mindful yoga, insight meditation, walk meditation), sharing of experiences of these exercises, reflections in small groups, psycho-education (e.g., stress, depression, self-care), and review of home practices. An overview of core elements is given in Van der Gucht et al. (2017b).
  The MBI is supported by homework assignments and audio material. Groups will include 5 participants, yielding 6 groups in total. The MBI will be delivered by highly qualified certified trainers with more than 10 years of experience in mindfulness meditation and extensive experience working with adolescents. Trainers will attend inter- and supervision moments on a regular basis to check treatment fidelity and trainer adherence.

SUMMARY:
Adolescents with chronic conditions often experience high levels of stress, anxiety and depression and reduced quality of life. Mindfulness-Based Interventions (MBI) have been found to improve emotional distress in clinical and non-clinical populations. Recent reviews suggest that MBIs are a promising technique to support adolescents with a chronic condition in managing their symptoms and ultimately enhance their quality of life.

To test the effects of an MBI on emotional distress and quality of life and delineate the underlying mechanisms, the You.Mind! study uses a randomised staggered within-subjects design. 30 adolescents with a chronic condition (taking drop-out into account) will be randomised to a baseline phase of 14 to 28 days followed by an MBI, consisting of 4 online group sessions and online support spread over 8 weeks. Outcomes will be assessed by short, repeated measurements throughout the baseline, training, and follow-up phases and by standardized questionnaires and experience sampling measures before randomisation, at post-intervention and 3-months follow-up. Analysis will be based on general linear modelling and multilevel mixed-effects modelling. The investigators hypothesize that a MBI can help adolescents with a chronic condition to reduce their symptoms of stress, anxiety and depression, and increase their quality of life.

DETAILED DESCRIPTION:
Once a pool of 15 participants has been enrolled, they will be randomised to one of three MBI groups, which start their training with half a week time lag. Within each group, participants will be randomised to a baseline phase of 2, 2.5, 3, 3.5 or 4 weeks, with 3-4 days between starting points of individual participants. Thus, the baseline phase will start at different time points for participants within the same group to enable them to start the intervention simultaneously while having baseline phases of varying length. Participants from different groups may begin their baseline phase at the same time while their intervention starts at a different time point. The same procedure will be repeated for the second pool of 15 participants.

ELIGIBILITY:
Inclusion Criteria:

* The adolescents suffer from a chronic condition lasting one year or more that impairs functional mobility and/or requires ongoing medical care.
* They should understand and speak Dutch.
* Written informed consent (including informed consent from a parent for those <18yrs) after having been informed on all aspects of the study.

Exclusion Criteria:

* Evidence of a current or lifetime severe mental illness.
* Current treatment for a psychiatric disorder.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Distress | Before the baseline phase (pre-measurement), during the baseline phase, during the intervention phase, in the week after the intervention (post-measurement), during the follow-up phase, and 3 months after the intervention (follow-up measurement)
  A 3-item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to measure feelings of anxiety, stress and depression in the present moment. The same scale is used for all other visual analogue scales.
Change in Pediatric Quality of Life InventoryTM (PedsQLTM 4.0; Varni, Seid & Kurtin, 2001) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The PedsQLTM is a 23-item scale designed to assess four domains of health, namely physical functioning, emotional functioning, social functioning, and school functioning in adolescents in the past month. Items are scores on a 5-point Likert scale ranging from "0" (never) to "4" (almost always).

SECONDARY OUTCOMES:
Change in the Depression Anxiety Stress Scales (DASS-21; Lovibond & Lovibond, 1995) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The DASS is a 21-item scale and is comprised of three sub-scales that measure symptoms of depression, anxiety and stress over the past week. Items are scored on a 4-point Likert scale ranging from "0" (did not apply to me at all) to "3" (applied to me very much or most of the time).
Change in the Leuven Anhedonia Self-report Scale (LASS; Bastin, Nelis, Raes, Vasey, & Bijttebier, 2018) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The LASS is a 12-item scale designed to assess consummatory, anticipatory, and motivational aspects of anhedonia over the past two weeks. Items are scored on a 5-point Likert scale ranging from "1" (completely untrue) to "5" (completely true).
Change in the Dampening subscale of Responses to Positive Affect questionnaire (RPA; Feldman, Joormann, & Johnson, 2008) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The dampening subscale of the RPA is used to measure dampening responses to positive affective states using 6 items on a 4-point Likert scale ranging from "1"(almost never) to "4"(almost always).
Change in the Non-Acceptance and Suppression of Negative Emotions Scale (NASNES) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The NASNES is a 10-item scale designed to assess the extent of suppression vs. acceptance of negative emotions on a 7-point Likert scale ranging from "1"(not at all) to "7"(very much).
Change in the Core Characteristics Subscale of the Perseverative Thinking Questionnaire (PTQ; Ehring et al., 2011) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The core characteristics subscale of the PTQ measures the main characteristics of repetitive negative thinking, namely the repetitiveness, the intrusiveness and the difficulty of disengaging. Its 9 items are rated on a 5-point Likert scale ranging from "0" (never) to "4" (always).
Change in the Self-Compassion Scale - Short Form (SCS-SF; Raes, Pommier, Neff, & van Gucht, 2011) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The 12-item short form of the Self-Compassion Scale assesses the main components of self-compassion, namely self-kindness vs. self-judgment, common humanity vs. isolation and mindfulness vs. over-identification. Items are rated on a 5-point Likert scale ranging from "1" (almost never) to "5" (almost always).
Change in the Short Form of the Comprehensive Inventory of Mindfulness Experiences (CHIME-SF; Johnson, Burke, Brinkman, & Wade, 2017) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The 24-item CHIME-SF measures different mindfulness skills including awareness of internal experiences, awareness of external experiences, acting with awareness, accepting and non-judgmental attitude, nonreactive decentering, openness to experiences, awareness of thought's relativity, and insightful understanding using a 6-point Likert scale ranging from "1" (almost never) to "6" (almost always).
Change in adapted version of Pain Solutions Questionnaire (PaSol; de Vlieger, van den Bussche, Eccleston, & Crombez, 2006) | Before the baseline phase (pre-measurement), in the week after the intervention (post-measurement) and 3 months after the intervention (follow-up)
  The 14-item adapted PaSol scale is used to measure participants' acceptance of their illness/condition on a 7-point Likert scale ranging from "1" (not at all) to "6" (very much).
Change in (Non)Acceptance of Negative Emotions | Before the baseline phase (pre-measurement), during the baseline phase, during the intervention phase, in the week after the intervention (post-measurement), during the follow-up phase, and 3 months after the intervention (follow-up measurement)
  A 2-item visual analogue scale assesses the acceptance and non-acceptance of negative emotions since the last beep.
Change in Anhedonia | Before the baseline phase (pre-measurement), during the baseline phase, during the intervention phase, in the week after the intervention (post-measurement), during the follow-up phase, and 3 months after the intervention (follow-up measurement)
  A 3-item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" measures aspects of anhedonia in the present moment. The final score will be computed as the average of the individual items.
Change in Dampening | Before the baseline phase (pre-measurement), during the baseline phase, during the intervention phase, in the week after the intervention (post-measurement), during the follow-up phase, and 3 months after the intervention (follow-up measurement)
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to assess dampening of positive emotions since the last beep.
Change in Repetitive Negative Thinking (RNT) - worry | Before the baseline phase (pre-measurement), during the baseline phase, during the intervention phase, in the week after the intervention (post-measurement), during the follow-up phase, and 3 months after the intervention (follow-up measurement)
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" is used to measure worry since the last beep.
Change in Self-compassion | Before the baseline phase (pre-measurement), during the baseline phase, during the intervention phase, in the week after the intervention (post-measurement), during the follow-up phase, and 3 months after the intervention (follow-up measurement)
  A single item visual analogue scale ranging from 0 to 100 with the anchors "not at all" and "very much" measures self-compassion since the last beep.

OTHER OUTCOMES:
Harms and Unpleasant Experiences Survey (HUES) | In the week after the intervention (post-measurement)
  The HUES is designed to assess unpleasant and negative effects following mindfulness practice. Its 10 items are a combination of open-ended questions and closed-ended questions rated on different Likert scales.
Positive and negative aspects of mindfulness | 3 months after the intervention (follow-up)
  For open-ended assessment of difficulties and strengths of the MBI, participants will describe three positive and three negative aspects of their mindfulness meditation practice.

CONTACTS AND LOCATIONS:
Overall Officials: Katleen Van der Gucht, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Moderately sensitive information including age, demographic data, all other data coming from questionnaires and experience sampling data using smartphones will be pseudo-anonymized and shared upon reasonable request. To gain access, contact the authors at merle.kock@kuleuven.be (ORCID ID 0000-0001-9429-6321). The study protocol, statistical analysis plan and statistical code will be uploaded on clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The coded, pseudonomized dataset and supporting information (see above) will be available beginning from 3 months and ending 5 years after publication of the research results.
Access Criteria: Coded, pseudonomized data can be shared with regulatory authorities, ethical committees, other parties that collaborate with the research team and will be shared, as mentioned above, upon reasonable request. Other researchers will only have access to the coded, pseudonomized data, and only if they agree with the confidentiality rules agreed upon within this study.

REFERENCES:
- [Background] Barlow JH, Ellard DR. The psychosocial well-being of children with chronic disease, their parents and siblings: an overview of the research evidence base. Child Care Health Dev. 2006 Jan;32(1):19-31. doi: 10.1111/j.1365-2214.2006.00591.x. PMID 16398788
- [Background] Bastin M, Nelis S, Raes F, Vasey MW, Bijttebier P. Party Pooper or Life of the Party: Dampening and Enhancing of Positive Affect in a Peer Context. J Abnorm Child Psychol. 2018 Feb;46(2):399-414. doi: 10.1007/s10802-017-0296-3. PMID 28391490
- [Background] De Vlieger P, Van den Bussche E, Eccleston C, Crombez G. Finding a solution to the problem of pain: conceptual formulation and the development of the Pain Solutions Questionnaire (PaSol). Pain. 2006 Aug;123(3):285-293. doi: 10.1016/j.pain.2006.03.005. Epub 2006 May 3. PMID 16675113
- [Background] Ehring T, Zetsche U, Weidacker K, Wahl K, Schonfeld S, Ehlers A. The Perseverative Thinking Questionnaire (PTQ): validation of a content-independent measure of repetitive negative thinking. J Behav Ther Exp Psychiatry. 2011 Jun;42(2):225-32. doi: 10.1016/j.jbtep.2010.12.003. Epub 2010 Dec 21. PMID 21315886
- [Background] Feldman GC, Joormann J, Johnson SL. Responses to Positive Affect: A Self-Report Measure of Rumination and Dampening. Cognit Ther Res. 2008 Aug 1;32(4):507-525. doi: 10.1007/s10608-006-9083-0. PMID 20360998
- [Background] Johnson C, Burke C, Brinkman S, Wade T. Development and validation of a multifactor mindfulness scale in youth: The Comprehensive Inventory of Mindfulness Experiences-Adolescents (CHIME-A). Psychol Assess. 2017 Mar;29(3):264-281. doi: 10.1037/pas0000342. Epub 2016 Jun 2. PMID 27254018
- [Background] Kabat-Zinn J. Full catastrophe living: How to cope with stress, pain and illness using mindful meditation. New York: Delacorte. 1990.
- [Background] Lovibond SH, Lovibond PF. Manual for the depression anxiety stress scales. Psychology Foundation of Australia. 1996.
- [Background] Pinquart M, Shen Y. Depressive symptoms in children and adolescents with chronic physical illness: an updated meta-analysis. J Pediatr Psychol. 2011 May;36(4):375-84. doi: 10.1093/jpepsy/jsq104. Epub 2010 Nov 18. PMID 21088072
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Santos T, de Matos MG, Simoes C, Leal I, do Ceu Machado M. (Health-related) quality of life and psychosocial factors in adolescents with chronic disease: a systematic literature review. Int J Adolesc Med Health. 2017 Nov 23;31(4). doi: 10.1515/ijamh-2017-0037. PMID 29168956
- [Background] Segal ZV, Williams JMG. Mindfulness-Based Cognitive Therapy for Depression: A New Approach to Preventing Relapse (2nd ed.). New York: Guilford Publications Inc. 2012.
- [Background] Van der Gucht K, Takano K, Kuppens P, Raes F. Potential Moderators of the Effects of a School-Based Mindfulness Program on Symptoms of Depression in Adolescents. Mindfulness. 2017; 8(3): 797-806. https://doi.org/10.1007/s12671-016-0658-x
- [Background] Van der Gucht K, Takano K, Labarque V, Vandenabeele K, Nolf N, Kuylen S, Cosyns V, Van Broeck N, Kuppens P, Raes F. A Mindfulness-Based Intervention for Adolescents and Young Adults After Cancer Treatment: Effects on Quality of Life, Emotional Distress, and Cognitive Vulnerability. J Adolesc Young Adult Oncol. 2017 Jun;6(2):307-317. doi: 10.1089/jayao.2016.0070. Epub 2016 Dec 21. PMID 28002681
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Abujaradeh H, Safadi R, Sereika SM, Kahle CT, Cohen SM. Mindfulness-Based Interventions Among Adolescents With Chronic Diseases in Clinical Settings: A Systematic Review. J Pediatr Health Care. 2018 Sep-Oct;32(5):455-472. doi: 10.1016/j.pedhc.2018.04.001. Epub 2018 Jun 22. PMID 29941236
- [Background] Ahola Kohut S, Stinson J, Davies-Chalmers C, Ruskin D, van Wyk M. Mindfulness-Based Interventions in Clinical Samples of Adolescents with Chronic Illness: A Systematic Review. J Altern Complement Med. 2017 Aug;23(8):581-589. doi: 10.1089/acm.2016.0316. Epub 2017 Mar 29. PMID 28355082
- [Background] Blanck P, Perleth S, Heidenreich T, Kroger P, Ditzen B, Bents H, Mander J. Effects of mindfulness exercises as stand-alone intervention on symptoms of anxiety and depression: Systematic review and meta-analysis. Behav Res Ther. 2018 Mar;102:25-35. doi: 10.1016/j.brat.2017.12.002. Epub 2017 Dec 20. PMID 29291584
- [Background] Xunlin NG, Lau Y, Klainin-Yobas P. The effectiveness of mindfulness-based interventions among cancer patients and survivors: a systematic review and meta-analysis. Support Care Cancer. 2020 Apr;28(4):1563-1578. doi: 10.1007/s00520-019-05219-9. Epub 2019 Dec 13. PMID 31834518
- [Background] Greeson JM, Chin GR. Mindfulness and physical disease: a concise review. Curr Opin Psychol. 2019 Aug;28:204-210. doi: 10.1016/j.copsyc.2018.12.014. Epub 2018 Dec 27. PMID 30785067
- [Background] Greeson JM, Zarrin H, Smoski MJ, Brantley JG, Lynch TR, Webber DM, Hall MH, Suarez EC, Wolever RQ. Mindfulness Meditation Targets Transdiagnostic Symptoms Implicated in Stress-Related Disorders: Understanding Relationships between Changes in Mindfulness, Sleep Quality, and Physical Symptoms. Evid Based Complement Alternat Med. 2018 May 13;2018:4505191. doi: 10.1155/2018/4505191. eCollection 2018. PMID 29861769
- [Background] Hofmann SG, Gomez AF. Mindfulness-Based Interventions for Anxiety and Depression. Psychiatr Clin North Am. 2017 Dec;40(4):739-749. doi: 10.1016/j.psc.2017.08.008. Epub 2017 Sep 18. PMID 29080597
- [Derived] Kock M, Van Hoecke E, Raes F, Van der Gucht K. Study protocol for You.Mind!: boosting first-line mental health care for YOUngsters suffering from chronic conditions with mindfulness: a randomised staggered within-subjects design. BMJ Open. 2021 Apr 9;11(4):e042648. doi: 10.1136/bmjopen-2020-042648. PMID 33837097